CLINICAL TRIAL: NCT03739333
Title: Early Diagnosis of Pseudoprogression Using 11C-Methionine PET-MRI After Concomitant Radiochemotherapy Treatment for Glioblastoma.
Acronym: TIGRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL18_0265; 2018-002016-27 (EudraCT Number)
Record Dates: First submitted 2018-11-06; First posted 2018-11-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Glioblastoma
Keywords: glioblastoma; 11C-Methionine PET-MRI; sensitivity; temozolomide; radiotherapy
MeSH Terms: conditions — Glioblastoma; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with glioblastoma (Experimental): implementation of 11C-Methionine PET-MRI
  Interventions: Other: 11C-Methionine PET-MRI

INTERVENTIONS:
Other: 11C-Methionine PET-MRI — Implementation 11C-Methionine PET-MRI performed for each patient in one place (department of nuclear medicine of Hospices Civils de Lyon). The 11C-Methionine PET-MRI will be performed after radiochemotherapy in patients with MRI suspicious of pseudoprogression.

SUMMARY:
Pseudoprogression is a phenomenon related to post-treatment rearrangements (including radiation necrosis). It appears early in the first year after treatment and accounts for 30 to 50% of patients followed with glioblastoma. On MRI (current gold standard with international therapeutic response evaluation criteria RANO 2010), pseudoprogression is manifested by a progression of morphological abnormalities (contrast enhancement, FLAIR hypersignal) and can simulate tumor recurrence, even though the corticosteroid improved or kept clinical symptoms stabilized. In view of prognosis, the current diagnostic tools have not enough diagnosis accuracy for differentiation between pseudo-progression and early tumor recurrence, and are based on MRI retrospective analysis (2-3 months after). Recurrence of glioblastoma, is characterized by a higher amino acid metabolism than pseudoprogression, also 11C-Methionine (11C-MET), positron emitting radiotracer, showed promising results to differentiate these two entities. To date, hybrid 11C-MET PET-MRI studies remains limited to small sample size (a few dozen patients), and none focuses exclusively on glioblastoma.

Hypothesis of our study is that 11C-MET PET-MRI may be performed as a first-line MRI for suspected pseudoprogression and may changes therapeutic decision making and also patient prognosis.

The main objective is to evaluate the performance of hybrid PET-MRI imaging with 11C-MET to differentiate pseudoprogression from glioblastoma recurrence in patients treated with surgery and radiochemotherapy, compared to multimodality MRI).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or over,
* Patient with glioblastoma treated by radiochemotherapy with temozolomide,
* Patient with suspicion of pseudoprogression between the 1st and 12th month after the end of concomitant chemoradiotherapy,
* Patient receiving a social security scheme,
* Patient for whom informed and written consent to participate has been obtained,

Exclusion Criteria:

* Subject under safeguard of justice (tutelage, curatorship),
* Minor patient,
* Patient without signs of progression MRI (stable disease or good response to treatment according to the RANO 2010 criteria),
* Clinical or radiological progression justifying a change of treatment,
* Patient not able to decide and with refusal of the family entitled to continue research.
* Pregnant woman, breastfeeding or old enough to have children but without effective contraception,
* Contraindication to performing an MRI: permanently fixed metal parts (pacemaker, cerebral clip, cochlear implant, pin or screw for recent bone fracture, dental equipment, metal splinters), claustrophobia,
* Contraindication to gadolinium according to ANSM 2017 recommendations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-02-26 (Estimated); Study Completion 2025-01-26 (Estimated)

PRIMARY OUTCOMES:
false negatives and false positives description (diagnosis accuracy) of 11C-Methionine PET-MRI | within 1 months and 12 months post-treatment
  diagnosis accuracy of 11C-MET PET-MRI to differentiated pseudoprogression from tumor recurrence, compared to MRI. The gold-standard being retrospective MRI analysis.

SECONDARY OUTCOMES:
ROC curves for comparison of two diagnostic tests: MRI and PET-MRI | within 1 months and 24 months after inclusion
  use of area under the curve for each tests to identify the best
The proportion of pseudoprogression identified by PET-MRI to 11C-MET according to the genetic data | during 24 months after inclusion
  The proportion of pseudoprogression identified by PET-MRI to 11C-MET according to the methylation status of the O6-methylguanine-DNA- methyltransferase (MGMT) promoter, the level of expression of isocitrate dehydrogenase (IDH) mutation, ki67 and 1p19q mutation.
Overall survival analysis | during 24 months after inclusion
  Patients will be followed regularly for 2 years to assess overall survival at 12 months and at 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: DUCRAY François, Principal Investigator — Hospîces Civils de Lyon
Locations (1):
- Hopices Civils de Lyon, Bron, France